CLINICAL TRIAL: NCT01243645
Title: MP-1 Biofeedback: Pattern Stimulus Versus Audio-feedback in Age Related Macular Degeneration (AMD)
Brief Title: MP-1 Biofeedback: Pattern Stimulus Versus Audio-feedback in AMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Other Study IDs: BIO0110
Record Dates: First submitted 2010-11-17; First posted 2010-11-18 (Estimated); Last update posted 2010-11-18 (Estimated); Status verified 2010-09

CONDITIONS: Age Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: biofeedback training

SUMMARY:
Background:

Biofeedback techniques have demonstrated their uselfulness in the treatment of maculopathies. We wanted to evaluate the efficacy of visual rehabilitation by means of two different types of biofeedback techniques in patients with age related macular degeneration (AMD).

Methods:

30 patients bilaterally affected by AMD were enrolled with a mean age of 76,38±8,77 yrs. Patients were randomly divided in two groups: Group A was treated with an acoustic biofeedback, Group B with luminous biofeedback of a black and white checkerboard flickering during the examination. All patients underwent a complete ophthalmological examination. Rehabilitation consisted in 12 training sessions of 10 minutes for each eye performed once a week for both groups. Statistical analysis was performed using t- test. P values less than 0.05 were considered statistically significant.

Results:

Group A: visual acuity at the end of rehabilitation had improved, but this result was not statistically significant (p=0.054), reading speed showed a significant statistical improvement (p=0.031), as well as the fixation stability (p=0.0023) and single point mean retinal sensitivity value (p=0.044).

Group B: visual acuity improvement at the end of rehabilitation was statistically significant (p=0.048), reading speed showed a statistically significant improvement (p=0.024), as well as fixation stability (p=0.0012) and mean single point retinal sensitivity value (p=0.027). Final results for both groups were compared and patients in group B showed results which were statistically more significant.

Conclusion:

A contrast rich flickering biofeedback stimulus showed a statistically significant improvement in training the patients to modify their preferred retinal locus (PRL) in comparison to acoustic biofeedback. It is possible that increased involvement of the various retinal cell populations with visual stimuli create more efficient ganglion cell response that better utilize the residual retinal function.

ELIGIBILITY:
Inclusion Criteria:

* We enrolled 30 patients (18 women and 12 men), ranging in age from 56-89 with a mean of 76.38 ±8.77, bilaterally affected by neovascular AMD from the Medical Retina Unit of the Department of Ophthalmology, University La Sapienza of Rome, Polo Pontino, A. Fiorini Hospital from August 2009 to July 2010.

Diagnosis of neovascular AMD was based on a complete ophthalmological examination including anterior and posterior segment biomicroscopy, Fluorescein Angiography (Heidelberg HRA2 FA module Heidelberg Germany), spectral domain OCT (Heidelberg HRA-2 OCT module Heidelberg Germany), microperimetry with MP-1 (NIDEK Technologies Padua Italy).

Exclusion Criteria:

* Patients with other eye diseases (i.e. glaucoma, myopia, retinal detachment, etc), uncooperative patients and patients with media opacities were excluded.

Ages: 56 Years to 89 Years | Sex: All
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
improvement of visual acuity

SECONDARY OUTCOMES:
improvement of retinal sensitivity

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - University La Sapienza, Latina
  - Rome. Latina

REFERENCES:
- [Derived] Vingolo EM, Salvatore S, Limoli PG. MP-1 biofeedback: luminous pattern stimulus versus acoustic biofeedback in age related macular degeneration (AMD). Appl Psychophysiol Biofeedback. 2013 Mar;38(1):11-6. doi: 10.1007/s10484-012-9203-4. PMID 22903517